CLINICAL TRIAL: NCT04313608
Title: A Phase Ib, Open-Label, Multicenter Study Evaluating the Safety and Efficacy of Glofitamab or Mosunetuzumab in Combination With Gemcitabine Plus Oxaliplatin in Patients With Relapsed or Refractory Diffuse Large B-Cell Lymphoma and High-Grade Large B-Cell Lymphoma
Brief Title: A Study Evaluating the Safety and Efficacy of Glofitamab or Mosunetuzumab in Combination With Gemcitabine Plus Oxaliplatin in Participants With Relapsed or Refractory Diffuse Large B-Cell Lymphoma and High-Grade Large B-Cell Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GO41943
Record Dates: First submitted 2020-03-17; First posted 2020-03-18 (Actual); Results first posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2023-09

CONDITIONS: B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — glofitamab; Gemcitabine; Oxaliplatin; obinutuzumab; tocilizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Glofit-GemOx (Experimental): Participants will receive up to 8 cycles of Glofit-GemOx (glofitamab in combination with gemcitabine and oxaliplatin) administered in 21-day cycles, followed by up to 4 cycles of glofitamab monotherapy. A single dose of obinutuzumab will be administered 7 days prior to the first dose of glofitamab.
  Interventions: Drug: Glofitamab; Drug: Gemcitabine; Drug: Oxaliplatin; Drug: Obinutuzumab; Drug: Tocilizumab
- Arm B: Mosun-GemOx (Experimental): Participants will receive up to 8 cycles of Mosun-GemOx (mosunetuzumab in combination with gemcitabine and oxaliplatin) administered in 21-day cycles.
  Interventions: Drug: Gemcitabine; Drug: Oxaliplatin; Drug: Mosunetuzumab; Drug: Tocilizumab

INTERVENTIONS:
Drug: Glofitamab — Participants will receive intravenous (IV) glofitamab in combination with gemcitabine and oxaliplatin for up to 8 cycles, followed by up to 4 cycles of glofitamab monotherapy.
  Other Names: RO7082859
  Arms: Arm A: Glofit-GemOx
Drug: Gemcitabine — Participants will receive IV gemcitabine prior to oxaliplatin administration for up to 8 cycles.
Drug: Oxaliplatin — Participants will receive IV oxaliplatin after gemcitabine administration for up to 8 cycles.
Drug: Mosunetuzumab — Participants will receive IV mosunetuzumab in combination with gemcitabine and oxaliplatin for up to 8 cycles.
  Other Names: RO7030816
  Arms: Arm B: Mosun-GemOx
Drug: Obinutuzumab — Participants will receive a single dose of IV obinutuzumab 7 days prior to the first administration of glofitamab.
  Other Names: RO5072759
  Arms: Arm A: Glofit-GemOx
Drug: Tocilizumab — Participants will receive IV tocilizumab as needed to treat cytokine release syndrome (CRS).
  Other Names: RO4877533

SUMMARY:
This study is designed to evaluate the safety and efficacy of glofitamab or mosunetuzumab in combination with gemcitabine and oxaliplatin (Glofit-GemOx or Mosun-GemOx) in participants with relapsed or refractory (R/R) diffuse large B-cell lymphoma (DLBCL) or high-grade B-cell lymphoma (HGBCL).

ELIGIBILITY:
Inclusion Criteria

* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0,1, or 2
* Histologically confirmed B-cell lymphoma, including one of the following diagnoses per the 2016 World Health Organization (WHO) classification of lymphoid neoplasms: DLBCL, not otherwise specified (NOS); HGBCL with MYC and BCL2 and/or BCL6 rearrangements; HGBCL, NOS
* R/R disease, defined as follows: Relapse: disease that has recurred following a response that lasted >/=6 months after completion of last line of therapy; Refractory: disease that progressed during therapy or progressed within 6 months (<6 months) of prior therapy
* At least one line of prior systemic therapy
* At least one bi-dimensionally measurable nodal lesion or one bi-dimensionally measurable extranodal lesion, as measured on positron emission tomography-computed tomography (PET/CT) scan
* Adequate hematologic function
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods, and agreement to refrain from donating eggs, as follows: Women must remain abstinent or use contraceptive methods with a failure rate of <1% per year during the treatment period and for at least 18 months after the final dose of obinutuzumab, 6 months after the final dose of gemcitabine, 9 months after the final dose of oxaliplatin, 3 months after the final dose of mosunetuzumab, 3 months after the final dose of tocilizumab, and 2 months after the final dose of glofitamab. Women must refrain from donating eggs during this same period
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods, and agreement to refrain from donating sperm, as follows: With a female partner of childbearing potential or pregnant female partners, men must remain abstinent or use a condom plus an additional contraceptive method that together result in a failure rate of <1% per year during the treatment period and for at least 2 months after the final dose of glofitamab, 2 months after the final dose of mosunetuzumab, 2 months after the final dose of tocilizumab (if applicable), 3 months after the final dose of obinutuzumab, and 6 months after the final dose of oxaliplatin or gemcitabine to avoid exposing the embryo. Men must refrain from donating sperm during this same period.

Exclusion Criteria

* Participant has failed only one prior line of therapy and is a candidate for stem cell transplantation
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies (or recombinant antibody-related fusion proteins) or known sensitivity or allergy to murine products
* Contraindication to obinutuzumab, gemcitabine, oxaliplatin, or tocilizumab
* Prior treatment with a bispecific antibody targeting both CD20 and CD3, including glofitamab and mosunetuzumab
* Grade >1 peripheral neuropathy
* Treatment with radiotherapy, chemotherapy, immunotherapy, immunosuppressive therapy, or any investigational agent for the purposes of treating cancer within 2 weeks prior to first study treatment
* Treatment with monoclonal antibodies for the purposes of treating cancer within 4 weeks prior to the first study treatment
* Primary or secondary central nervous system (CNS) lymphoma at the time of recruitment or history of CNS lymphoma
* Current or history of CNS disease, such as stroke, epilepsy, CNS vasculitis, or neurodegenerative disease
* History of other malignancy that could affect compliance with the protocol or interpretation of results
* Evidence of significant, uncontrolled concomitant diseases that could affect compliance with the protocol or interpretation of results, including significant cardiovascular disease (such as New York Heart Association Class III or IV cardiac disease, myocardial infarction within the last 6 months, unstable arrhythmias, or unstable angina) or significant pulmonary disease (including obstructive pulmonary disease and history of bronchospasm)
* Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) at study enrollment or any major episode of infection (as evaluated by the investigator) within 4 weeks prior to first study treatment
* Suspected or latent tuberculosis
* Positive test results for chronic hepatitis B virus (HBV) infection
* Positive test results for hepatitis C virus (HCV) antibody
* Known HIV-seropositive status
* Known or suspected chronic active Epstein-Barr virus infection
* Known or suspected history of hemophagocytic lymphohistiocytosis (HLH)
* History of progressive multifocal leukoencephalopathy
* Adverse events from prior anti-cancer therapy that have not resolved to Grade 1 or better (with the exception of alopecia and anorexia)
* Administration of a live, attenuated vaccine within 4 weeks prior to the first study treatment administration or anticipation that such a live, attenuated vaccine will be required during the study
* Prior solid organ transplantation
* Prior allogenic stem cell transplant
* Active autoimmune disease requiring treatment
* Prior treatment with systemic immunosuppressive medications (including, but not limited to, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor agents) within 4 weeks prior to the first dose of study treatment
* Corticosteroid therapy within 2 weeks prior to first dose of study treatment, with exceptions defined by the study protocol
* Recent major surgery (within 4 weeks before the first study treatment) other than for diagnosis
* Clinically significant history of liver disease, including cirrhosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2020-06-04 (Actual); Primary Completion 2021-10-26 (Actual); Study Completion 2021-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (3):
- Australia (3):
  - Prince of Wales Hospital; Haematology, Randwick, New South Wales
  - Monash Health Monash Medical Centre, Clayton, Victoria
  - St Vincent's Hospital Melbourne, Fitzroy, Victoria

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: Glofit-GemOx: Participants received a single IV dose of obinutuzumab 7 days prior to their first dose of glofitamab. Participants then received up to 8 cycles of glofitamab + gemcitabine + oxaliplatin, followed by up to 4 additional cycles of glofitamab monotherapy (cycle length = 21 days)
- Arm B: Mosun-GemOx: Participants received up to 8 cycles of mosunetuzumab + gemcitabine + oxaliplatin (cycle length = 21 days)
Period: Overall Study
Arm/Group | Arm A: Glofit-GemOx | Arm B: Mosun-GemOx
Started | 17 | 6
Completed | 5 | 3
Not Completed | 12 | 3
Not completed — Death | 12 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Glofit-GemOx | Arm B: Mosun-GemOx | Total
Number analyzed (Participants) | 17 | 6 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.1 (8.7) | 69.3 (18.3) | 63.3 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 13 | 4 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 17 | 6 | 23
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 15 | 5 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Deaths Due to Adverse Events (AEs)
Description: An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Pre-existing conditions which worsen during a study are also considered as adverse events.
Time Frame: Baseline - 90 days after last dose of study treatment
Measure: Number; unit: Participants
Groups:
- Arm A: Glofit-GemOx: Participants received a single intravenous (IV) dose of obinutuzumab 7 days prior to their first dose of glofitamab. Participants then received up to 8 cycles of glofitamab + gemcitabine + oxaliplatin, followed by up to 4 additional cycles of glofitamab monotherapy (cycle length = 21 days).
Arm/Group | Arm A: Glofit-GemOx | Arm B: Mosun-GemOx
Number analyzed (Participants) | 17 | 6
Participants | 1 | 0

2. Secondary Outcome: Tolerability of Study Treatment as Measured by Dose Interruptions, Dose Reductions, and Treatment Discontinuation Due to AEs
Time Frame: Up to approximately 16 months
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: Glofit-GemOx | Arm B: Mosun-GemOx
Number analyzed (Participants) | 17 | 6
percentage of participants
  AEs leading to treatment discontinuation | 5.9 | 16.7
  AEs leading to dose modification or interruption | 29.4 | 50.0

3. Secondary Outcome: Complete Response (CR) Based on PET/CT as Determined by the Investigator According to the 2014 Lugano Response Criteria
Description: Per the 2014 Lugano Response Criteria for malignant lymphoma a CR = complete metabolic response with a score of 1, 2, or 3 on a 5-point scale (5PS), with higher scores indicating more extensive disease.
Time Frame: Up to approximately 16 months
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Arm A: Glofit-GemOx | Arm B: Mosun-GemOx
Number analyzed (Participants) | 17 | 6
percentage | 23.5 [6.81 to 49.90] | 50.0 [11.81 to 88.19]

4. Secondary Outcome: Objective Response Rate (ORR), Defined as the Proportion of Participants With a Best Overall Response of Partial Response (PR) or CR, as Determined by the Investigator According to the 2014 Lugano Response Criteria
Description: Per the 2014 Lugano Response Criteria for malignant lymphoma a CR = complete metabolic response with a score of 1, 2, or 3 on a 5-point scale (5PS), while a PR = partial metabolic response with a score of 4 or 5 on 5PS with higher scores indicating more extensive disease.
Time Frame: Up to approximately 16 months
Measure: Number; unit: Proportion expressed as percentage
Arm/Group | Arm A: Glofit-GemOx | Arm B: Mosun-GemOx
Number analyzed (Participants) | 17 | 6
Proportion expressed as percentage | 35.3 | 50.0

5. Secondary Outcome: Maximum Serum Concentration (Cmax) of Glofitamab
Time Frame: Cycle 1 Day 8 and Cycle 2 Day 1
Population: The pharmacokinetic population consisted of all participants that received at least one dose of glofitamab or mosunetuzumab and who had data from at least one post-dose sample.
Measure: Median (Full Range); unit: ug/mL
Arm/Group | Arm A: Glofit-GemOx
Number analyzed (Participants) | 17
ug/mL
  Pre-infusion Cycle 1 Day 8: number analyzed (Participants) | 15
  Pre-infusion Cycle 1 Day 8 | 0 [0 to 0]
  Within 30 mins post infusion Cycle 1 Day 8: number analyzed (Participants) | 16
  Within 30 mins post infusion Cycle 1 Day 8 | 0.6 [0.3 to 1.7]
  12 hours post infusion Cycle 1 Day 8 | 0.6 [0.1 to 0.9]
  24 hours post infusion Cycle 1 Day 8 | 0.5 [0.1 to 0.8]
  48 hours post infusion Cycle 1 Day 8: number analyzed (Participants) | 7
  48 hours post infusion Cycle 1 Day 8 | 0.3 [0 to 0.4]
  Pre-infusion Cycle 2 Day 1: number analyzed (Participants) | 16
  Pre-infusion Cycle 2 Day 1 | 0.8 [0.1 to 1.3]
  Within 30 minutes post infusion Cycle 2 Day 1: number analyzed (Participants) | 16
  Within 30 minutes post infusion Cycle 2 Day 1 | 9 [6.8 to 17.7]
  6 hours post infusion Cycle 2 Day 1: number analyzed (Participants) | 15
  6 hours post infusion Cycle 2 Day 1 | 7.8 [5.5 to 13.1]
  20 hours post infusion Cycle 2 Day 1: number analyzed (Participants) | 16
  20 hours post infusion Cycle 2 Day 1 | 6.5 [4.4 to 11.2]
  44 hours post infusion Cycle 2 Day 1: number analyzed (Participants) | 2
  44 hours post infusion Cycle 2 Day 1 | 3.8 [3.2 to 4.3]

6. Primary Outcome: Number of Treatment Discontinuations Due to AE
Description: as for outcome 1
Time Frame: Baseline - 90 days after last dose of study treatment
Measure: Number; unit: Participants
Arm/Group | Arm A: Glofit-GemOx | Arm B: Mosun-GemOx
Number analyzed (Participants) | 17 | 6
Participants | 1 | 1

7. Primary Outcome: Proportion of Participants With Serious Adverse Events (SAEs)
Description: as for outcome 1
Time Frame: Baseline - 90 days after last dose of study treatment
Measure: Number; unit: Proportion expressed as percentage
Arm/Group | Arm A: Glofit-GemOx | Arm B: Mosun-GemOx
Number analyzed (Participants) | 17 | 6
Proportion expressed as percentage | 70.6 | 66.7

8. Primary Outcome: Proportion of Participants With Cytokine Release Syndrome (CRS) by Grade of Severity
Description: Severity of CRS was determined according to the American Society for Transplantation and Cell Therapy (ASTCT) Consensus Grading Criteria, in which Grade 1 as fever (≥38.0°C) with or without other symptoms; Grade 2 as fever with hypotension not requiring vasopressors and/or hypoxia requiring the use of oxygen (low-flow); and Grade 3 as fever with hypotension requiring one vasopressor with or without vasopressin and/or hypoxia requiring the use of oxygen (high-flow).
Time Frame: Baseline - 90 days after last dose of study treatment
Measure: Number; unit: Proportion expressed as percentage
Arm/Group | Arm A: Glofit-GemOx | Arm B: Mosun-GemOx
Number analyzed (Participants) | 17 | 6
Proportion expressed as percentage
  Grade 1 | 29.4 | 16.7
  Grade 2 | 11.8 | 0
  Grade 3 | 5.9 | 0

ADVERSE EVENTS:
Time Frame: Baseline - 90 days after the final dose of study treatment
Arm/Group | Arm A: Glofit-GemOx | Arm B: Mosun-GemOx
All-Cause Mortality (participants affected / at risk) | 1/17 | 0/6
Serious Adverse Events (participants affected / at risk) | 12/17 | 4/6
Other Adverse Events (participants affected / at risk) | 17/17 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Glofit-GemOx (N=17) | Arm B: Mosun-GemOx (N=6)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 6 (6) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 2 (4) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 3 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (2)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Immune effector cell-associated neurotoxicity syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Glofit-GemOx (N=17) | Arm B: Mosun-GemOx (N=6)
Anaemia (Blood and lymphatic system disorders) | 6 (15) | 3 (5)
Neutropenia (Blood and lymphatic system disorders) | 4 (5) | 1 (8)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (6) | 2 (4)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Blepharitis (Eye disorders) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal tenderness (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 4 (4) | 3 (4)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 5 (10)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (5) | 4 (5)
Oesophageal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 4 (4) | 4 (4)
Oedema peripheral (General disorders) | 0 (0) | 2 (3)
Performance status decreased (General disorders) | 1 (1) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 7 (14) | 0 (0)
Hypogammaglobulinaemia (Immune system disorders) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 2 (4)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1)
Cytomegalovirus infection reactivation (Infections and infestations) | 1 (1) | 0 (0)
External ear cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 3 (3) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (2) | 3 (5)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 2 (2) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0)
Liver function test abnormal (Investigations) | 4 (5) | 0 (0)
Neutrophil count decreased (Investigations) | 3 (4) | 0 (0)
Platelet count decreased (Investigations) | 4 (7) | 0 (0)
Weight decreased (Investigations) | 3 (3) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 2 (3)
Hypomagnesaemia (Metabolism and nutrition disorders) | 6 (9) | 4 (5)
Hypophosphataemia (Metabolism and nutrition disorders) | 4 (4) | 4 (9)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 1 (1)
Intention tremor (Nervous system disorders) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 3 (3) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 6 (7) | 1 (1)
Paraesthesia (Nervous system disorders) | 2 (2) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (4) | 3 (3)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Prostatomegaly (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Flushing (Vascular disorders) | 2 (5) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
Superficial vein thrombosis (Vascular disorders) | 2 (2) | 1 (2)
Thrombophlebitis (Vascular disorders) | 0 (0) | 2 (2)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Vasospasm (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-02): https://cdn.clinicaltrials.gov/large-docs/08/NCT04313608/Prot_SAP_000.pdf